CLINICAL TRIAL: NCT01827202
Title: Renin-Angiotensin-System Quantification in Patients Treated With Aliskiren or Candesartan (RASQAL)
Brief Title: RAS Quantification in Patients With Aliskiren or Candesartan
Acronym: RASQAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marcus Saemann, Assoc. Prof. Priv.-Doz. Dr.med.univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: EK-Nr. 011/2012
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Hypertension; Chronic Kidney Disease; Proteinuria
Keywords: renin-angiotensin-system; RAS blockade
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic; Proteinuria | interventions — aliskiren; candesartan; candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aliskiren (Active Comparator): After a two-week phase where all RAS blockade is eliminated, patients in this arm will commence taking aliskiren 150 mg once daily for 4 weeks. Thereafter, the dose will be increased to 300 mg once daily for another 4 weeks.
  Interventions: Other: RAS blockade discontinuation; Drug: Aliskiren
- Candesartan (Active Comparator): After a two-week phase where all RAS blockade is eliminated, patients in this arm will commence taking candesartan 8 mg once daily for 4 weeks. Thereafter, the dose will be increased to 16 mg once daily for another 4 weeks.
  Interventions: Other: RAS blockade discontinuation; Drug: Candesartan

INTERVENTIONS:
Other: RAS blockade discontinuation — In the initial two weeks of the study, all RAS blockade will be eliminated from the subjects' antihypertensive regimen
Drug: Aliskiren
  Other Names: Rasilez
  Arms: Aliskiren
Drug: Candesartan
  Other Names: Atacand
  Arms: Candesartan

SUMMARY:
Forced blockade of the renin-angiotensin-system (RAS) by using direct renin inhibition (DRI) has long been propagated to effectuate beneficial outcomes. However, recent large clinical trials have outlined harmful effects for DRI in combination with other forms of RAS blockade. To date, information regarding DRI as RAS-blocking monotherapy is very limited. Furthermore, it remains to be elucidated how DRI and angiotensin receptor blockers affect the so-called 'classical' and 'alternative' RAS molecularly. As components of the 'alternative' RAS (e.g. Ang 1-7) have moved into research focus, it would be of importance to determine angiotensin regulation with medical RAS blockade.

In this prospective, single-center randomized trial over 10 weeks, 24 patients with chronic kidney disease (CKD) stage III-IV (eGFR 15-59 ml/min) will be randomized to take either aliskiren (up to 300 mg per day) or candesartan (up to 16 mg per day) after a two week run-in phase where all RAS-blockers are eliminated. The investigators will then employ a novel mass spectrometry-based quantification method (after run-in and 10 weeks) to capture the concentrations of ten different angiotensin peptides (including angiotensin I and II, angiotensin 1-7 and angiotensin 1-5).

The investigators hypothesize that significant differences exist between angiotensin levels in CKD patients with DRI compared to angiotensin receptor blockers. Specifically, the investigators expect to determine the regulation of the alternative RAS represented by angiotensin 1-7 with proximal versus distal blockade of the system.

Our data might contribute to a more profound understanding of results from registries and clinical trials beyond the clinical effects of RAS blockade. Further, the study's results might help to individualize and optimize RAS-blocking therapy strategies in CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stages III-IV (defined by modification of diet in renal disease (MDRD) formula)
* Urinary albumin to creatinine ratio (UACR) >300mg/g, UACR >200mg/g if already receiving RAS blockade
* Arterial hypertension

Exclusion Criteria:

* Age <18 years
* Diabetes mellitus type 2 (defined by WHO criteria)
* Chronic kidney disease stage V (end-stage renal disease)
* UACR >3500mg/g
* Severe hypertension (systolic blood pressure >180mmHg)
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Mass spectrometry RAS peptide quantification | 2 months
  Quantitative RAS peptide changes determined by mass spectrometry after a 2-month treatment with aliskiren or candesartan

SECONDARY OUTCOMES:
Blood pressure | 2 months
  Blood pressure reduction, determined by ambulatory blood pressure measurements at study start and end
Proteinuria | 2 months
  Proteinuria reduction, measured by urinary albumin/creatinine ratio at study start and end

CONTACTS AND LOCATIONS:
Overall Officials: Marcus D Saemann, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Internal Medicine III, Division of Nephrology and Dialysis, Vienna, Vienna, Austria